CLINICAL TRIAL: NCT04115917
Title: Scleral Depression Pain With Schocket Depressor and Cotton Tipped Applicator: Depression Eye Pain Relief Evaluation Study (DEPRESS)
Brief Title: Evaluation of Discomfort Associated With Scleral Depression During Retina Examinations
Acronym: DEPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Joseph Raevis, Ophthalmologist, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: JJR666
Record Dates: First submitted 2019-09-21; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Retina--Diseases; Retinal Detachment; Retinal Degeneration
Keywords: Scleral Depression; Visual Analog Scale; Pain; Discomfort; Schocket Scleral Depressor; Cotton Tipped Applicator; Diabetes
MeSH Terms: conditions — Retinal Detachment; Retinal Degeneration; Pain; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The first eye to undergo scleral depression was randomly assigned, then that eye was randomized two either of the scleral depression methods. The contralateral eye then had the alternative method of scleral depression performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schocket Scleral Depressor (Experimental): Scleral Depression with Schocket Scleral Depressor
  Interventions: Device: Cotton tipped applicator
- Cotton Tipped Applicator (Active Comparator): Scleral Depression with Cotton Tipped Applicator
  Interventions: Device: Schocket scleral depressor

INTERVENTIONS:
Device: Schocket scleral depressor — Scleral Depression on eye with Schocket scleral depressor
  Arms: Cotton Tipped Applicator
Device: Cotton tipped applicator — Scleral Depression on eye with cotton tipped applicator
  Arms: Schocket Scleral Depressor

SUMMARY:
Scleral depression is an important technique used to examine the peripheral retina but often causes patient discomfort. The goal of this study was to compare levels of discomfort during scleral depression with a Schocket scleral depressor and cotton tipped applicator.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who received dilated eye examinations in the retina or general eye clinic

Exclusion Criteria:

* Younger than 18
* Pregnant
* Prior scleral buckle, filtering bleb or underwent any other ocular surgery within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Discomfort During Scleral Depression with Schocket Depressor and Cotton Tipped Applicator | Pain evaluated immediately scleral depression was completed on the eye
  Visual Analog Scale (VAS) was used to evaluate pain immediately after scleral depression was completed. The VAS scale used was a 100mm long line with 0 representing no pain at all and 100 representing the worst pain possible.

SECONDARY OUTCOMES:
Hemoglobin A1c | 1 year
  The association of discomfort experienced during scleral depression and the patients hemoglobin A1c.
Spherical Equivalent of Glasses Prescription | 1 day
  The association of discomfort experienced during scleral depression and the patients spherical equivalent of their glasses prescription.
Age | 1 day
  The association of discomfort experienced during scleral depression and the patients age based on those less than 65 versus those greater than 65 years of age
Left Eye vs Right Eye | 1 day
  The association of discomfort experienced during scleral depression and the patients left and right eyes. Of note, each eye had a separate method of scleral depression performed.
Retinal pathology | 1 day
  Discomfort during scleral depression in participants with peripheral retinal tears or holes versus patients with no peripheral retinal pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Raevis, MD, Principal Investigator — Kings County Hospital Department of Emergency Medicine
Locations (1):
- Kings County Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT04115917/Prot_SAP_000.pdf